CLINICAL TRIAL: NCT03942484
Title: Efficacy of Repetitive Pulse Magnetic Stimulation for Improvement of Urinary Incontinence and Female Sexual Function
Brief Title: Efficacy of rPMS for Improvement of Urinary Incontinence and Female Sexual Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: BTL Industries Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BTL-099-S
Record Dates: First submitted 2019-04-18; First posted 2019-05-08 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Urinary Incontinence
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment Group (Experimental): Treatment with the investigational device - rPMS
  Interventions: Device: rPMS device

INTERVENTIONS:
Device: rPMS device — Pelvic floor muscle contractions will be induced by the device.

SUMMARY:
Evaluation of the repetitive pulse magnetic stimulation (rPMS) for the treatment of urinary incontinence and a female sexual satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Age between 21 and 65 years
* Voluntarily signed informed consent form
* Suffers from UI
* Sexually active
* FSFI Questionnaire score ≤ 26.55 points

Exclusion Criteria:

* Suffers from other types of urinary incontinence other than SUI, UUI, MUI
* Currently lactating
* Cardiac pacemakers
* Implanted defibrillators and/or neurostimulators
* Electronic implants
* Metal implants, including copper IUD
* Drug pumps
* Hemorrhagic conditions
* Anticoagulation therapy
* Fever
* Pregnancy
* Following recent surgical procedures when muscle contraction may disrupt the healing process
* Application over areas of the skin which lack normal sensation

Ages: 21 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2019-05-01 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-10-20 (Actual)

PRIMARY OUTCOMES:
Evaluation of quality of life improvement using the ICIQ-UI questionnaire | 18 months
  Evaluation of change in ICIQ-UI score. Decrease of the score will be considered as an improvement.
Evaluation of quality of life improvement using the FSFI questionnaire | 18 months
  Evaluation of change in FSFI score. Increase of the score will be considered as an improvement.
Evaluation of quality of life improvement using the PISQ-12 questionnaire | 18 months
  Evaluation of change in PISQ-12 score. Increase of the score will be considered as an improvement.

SECONDARY OUTCOMES:
Safety evaluation: Incidence of adverse events (AE) associated with study device will be followed. | 18 months
  Incidence of adverse events (AE) associated with study device will be followed.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Julene Samuels, Louisville, Kentucky
  - Joseph Berenholz, Farmington Hills, Michigan
  - Gynecological Solutions, Hillsborough, New Jersey
  - Southern Urogynecology, West Columbia, South Carolina
  - Hillcroft Medical Clinic, Sugar Land, Texas